CLINICAL TRIAL: NCT06113770
Title: Clinical Evaluation of Polymethyl Methacrylate CAD/CAM Crowns Versus Prefabricated Zirconia Crowns in Primary Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Adel Sherif Mostafa Rehab (Other)
Responsible Party: Sponsor-Investigator, Adel Sherif Mostafa Rehab, Principal Investigator, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 787/4375
Record Dates: First submitted 2023-10-23; First posted 2023-11-02 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Caries of Infancy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ready made zirconia (Experimental): the selected tooth will receive ready made zirconia crown
  Interventions: Other: preparation of the tooth to receive ready made zirconia crown
- pmma crown (Experimental): the selected tooth will receive cad cam custom made pmma crown
  Interventions: Other: preparation of the tooth to receive CAD CAM PMMA custom made crown

INTERVENTIONS:
Other: preparation of the tooth to receive ready made zirconia crown — Occlusal reduction 1 to 2 mm using flame bur . Open the interproximal contacts. The tooth should be reduced circumferentially by approximately 0.5-1.5mm . The preparation margin should be carefully extended and refined to a feather-edge approximately 1-2mm subgingivally .
  Crown size will be determined using try in kit .
  Arms: ready made zirconia
Other: preparation of the tooth to receive CAD CAM PMMA custom made crown — * Open the interproximal contacts .
  * The tooth should be reduced circumferentially by approximately 0.5-1mm .
  * The preparation margin should be carefully extended and refined to a feather- edge approximately 1-2mm subgingivally .
  * Rubber base impression will be taken by BMS additional silicone kit to the prepared tooth and will be sent to the laboratory to be scanned and to design the crown .
  * The final crown will be cemented using glass ionomer cement .
  Arms: pmma crown

SUMMARY:
, in this studythe investigator will compare between ready-made zirconia crowns and Computer-aided design and Computer-aided manufacturing (CAD/CAM) polymethyl methacrylate (PMMA) crowns to overcome the disadvantages of ready-made zirconia crowns.

ELIGIBILITY:
A- Inclusion Criteria:

1. Primary molars indicated for crown restoration (pulp treated molars indicated for crown
2. Co-operative child (Frankel scale +ve and ++ve)
3. The age ranged from 4 to 8 years regardless of sex or socioeconomic background.

B- Exclusion Criteria:-

1. Badly decayed non-restorable tooth indicated for extraction.
2. Patients with parafunctional habits like bruxism.
3. Systemic diseases with oral manifestation or blood diseases.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 17 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Gingival condition | in 6 months
  Löe & Silness gingival index

SECONDARY OUTCOMES:
gingival bleeding | 6 months
  Papilla Bleeding Index

CONTACTS AND LOCATIONS:
Overall Officials: Adel S Rehab, Principal Investigator — Al-Azhar University
Locations (1):
- AlAzharU, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No